CLINICAL TRIAL: NCT01632475
Title: Long Term Follow-Up Study of the Safety and Exploratory Efficacy of Pneumostem® in Premature Infants With Bronchopulmonary Dysplasia
Brief Title: Follow-Up Study of Safety and Efficacy of Pneumostem® in Premature Infants With Bronchopulmonary Dysplasia
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Medipost Co Ltd. (Industry)
Responsible Party: Principal Investigator, Won Soon Park, Professor of Pediatrics, Samsung Medical Center
Other Study IDs: MP-CR-006-F/U
Record Dates: First submitted 2012-06-27; First posted 2012-07-03 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Human umbilical cord blood-derived mesenchymal stem cells; Premature infants; Bronchopulmonary dysplasia; Lung injury; Lung diseases; Hyperplasia; Ventilator-induced lung injury; Respiratory lung diseases; Pathologic Processes; Infant, Premature, Diseases; Infant, Newborn, Diseases
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Lung Injury; Lung Diseases; Hyperplasia; Ventilator-Induced Lung Injury; Pathologic Processes; Infant, Premature, Diseases; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pneumostem®: Low Dose Group (3 subjects): 1.0 x 10^7 cells/kg, High Dose Group (6 subjects): 2.0 x 10^7 cells/kg
  Interventions: Biological: Pneumostem®

INTERVENTIONS:
Biological: Pneumostem® — A single intratracheal administration
  Low Dose Group (3 patients): 1.0 x 10^7 cells/kg, High Dose Group (6 patients): 2 x 10^7 cells/kg
  * The subjects were administered with Pneumostem® in the earlier part of the phase I study. No drugs/biologics are administered during this part of the study.
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells

SUMMARY:
This is a long term follow-up study of the open label, single-center, phase I clinical trial to evaluate the safety of Pneumostem® in premature infants with BPD.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is the most common cause of death for premature newborns with low birth weights. In addition, many children who recover from the disease suffer from various complications such as prolonged hospitalization, pulmonary hypertension, and failure to thrive.

It has been reported that bone marrow-derived mesenchymal stem cells (BM-MSC) can differentiate into pulmonary epithelial and pulmonary endothelial cells. Some animal studies showed that BM-MSCs differentiate into bronchial cells and type 2 pneumocytes in rats with pneumonia and improve the fibrosis that occur after administration of bleomycin. Based on the findings, it is considered that mesenchymal stem cell therapy can help regenerate the damaged lung as well as BPD that cause lung inflammation, fibrosis, deficiency of type 2 pneumocytes, and so on.

PNEUMOSTEM® consists of human umbilical cord blood-derived mesenchymal stem cells and is intended to treat BPD in premature infants. This is a long term follow-up study of the earlier part of the phase I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* all Infants who enrolled in the Phase 1 PNEUMOSTEM® clinical trial (NCT01297205)

Exclusion Criteria:

* Infants whose parent or legal guardian did not want to participate in the study

Ages: 4 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who enrolled in the study of phase 1 clinical trial to evaluate the safety and efficacy of PNEUMOSTEM® Treatment in Premature Infants With Bronchopulmonary Dysplasia. (NCT01297205)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Adverse Drug Reaction | at corrected age of 21 months (±3 months)
  Blood test, chest x-ray, physical exam

SECONDARY OUTCOMES:
Neurological development test outcome from the subjects who were treated with Pneumostem®, compared with the patients who suffered from the same conditions but not treated with Pneumostem® | at corrected age of 10 months (±2 months) and 21 months (±3 months)
  Bayely test results of the 9 subjects who were treated with Pneumostem® during the early part of the Phase I study.
  The results of Brain MRI study performed at corrected age of 18-24 months.
Growth | Corrected gestational age of 4-6months, 8-12months, 18-24months
  Body weight, Head circumference, Height : growth percentile

CONTACTS AND LOCATIONS:
Overall Officials: Won-Soon Park, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ahn SY, Chang YS, Kim JH, Sung SI, Park WS. Two-Year Follow-Up Outcomes of Premature Infants Enrolled in the Phase I Trial of Mesenchymal Stem Cells Transplantation for Bronchopulmonary Dysplasia. J Pediatr. 2017 Jun;185:49-54.e2. doi: 10.1016/j.jpeds.2017.02.061. Epub 2017 Mar 21. PMID 28341525
- See also: Safety and Efficacy Evaluation of PNEUMOSTEM® Treatment in Premature Infants With Bronchopulmonary Dysplasia — http://clinicaltrials.gov/ct2/show/NCT01297205?term=pneumostem&rank=1